CLINICAL TRIAL: NCT04393272
Title: Digital Intelligent Assistant for Nursing Application Evaluation of 3-Dimensional Sensor Technology in Long Term Care and Acute Geriatrics. A Single Center Observational Study
Brief Title: Digital Intelligent Assistant for Nursing Application
Acronym: DIANA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Geriatrische Klinik St. Gallen (Other)
Responsible Party: Principal Investigator, Thomas Munzer, MD, PhD, Chief of Geriatrics, Geriatrische Klinik St. Gallen
Other Study IDs: BASEC 20-00904
Record Dates: First submitted 2020-05-11; First posted 2020-05-19 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Frailty Syndrome; Fall in Nursing Home; Dementia; Delirium in Old Age; Incontinence, Urinary; Incontinence Bowel
Keywords: 3D sensors; falls detection; toileting algorithm
MeSH Terms: conditions — Frailty; Dementia; Urinary Incontinence; Encopresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Three dimensional sensor system designed for fall detection (Fearless) — Detection of falls in nursing home residents and acute geriatric hospital patiients

SUMMARY:
This is an observational study that intends to compare falls or fall-risk related alarms derived from a three-dimensional sensor system with the clinical reality definded by attending nurses.

DETAILED DESCRIPTION:
Three dimensional sensor technology (3DS) is available for fall detection and fall prevention (e.g. unwanted getting up in persons with risks for frequent falls) in several institutions in Europe and Switzerland. 3DS are capable to analyze completely anonymized data and alert nurses towards a dangerous (fall) or potentially dangerous (getting out of bed) event during day- and nighttime. Multi-sensor technology has been applied to assess activities of daily living in persons cognitive problems living at home. To our knowledge, 3DS technology has not been examined as part of a structured clinical protocol. In addition, the combination of two digital technologies (3DS and a server based software) as an integrative platform could help to develop algorithms to analyze complex human activities such as using a toilet. Automated analyses of such complex activities have the potential to support nursing staff in the future.

ELIGIBILITY:
Inclusion criteria Informed consent given by person or caregiver Patients admitted

* with or without cognitive decline for any reason
* with acute and/or chronic conditions
* after any kind of surgery

Exclusion Criteria:

1. For Falls assessment by 3D sensors:

   • Based on the multifactorial risk for falls there are no exclusion criteria for falls assessment
2. For the development of toileting algorithm:

   * severe urine or fecal incontinence
   * permanent indwelling urinary catheter
   * permanent urinary or bowel stoma

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Due to the observationa design, we will have no control group. All persons admitted to the rooms equipped with this novel technology are asked to participate.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Falls detection rate | Through study completion, an average of 6 months
  Number of falls detected by the system compared to falls detected by nursing staff members

OTHER OUTCOMES:
Assessment of toileting | Through study completion, an average of 6 months
  3d sensor system data will be used to develop an algorithm for a complex activity such as using a toilet. The senors results will be compared with a Nurse led 12 step observation protocol. Parts of the activity model include: (1) enter the room, (2) go to the toilet, (3) take off clothes, (4) sit on the toilet, (5) clean oneself, (6) stand up, (7) get dressed, (8) flush the toilet, (9) go to the sink, (10) wash hands, (11) dry hands, (12) leave the room, as well as emergencies.

CONTACTS AND LOCATIONS:
Locations (1):
- Geriatrische Klinik, Sankt Gallen, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: No